CLINICAL TRIAL: NCT06485466
Title: Transarterial Chemoembolization Plus Camrelizumab and Apatinib for Unresectable Hepatocellular Carcinoma : a Randomised , Open Label, Multicenter Controlled Trial
Brief Title: TACE Plus Camrelizumab and Apatinib for Unresectable Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Guohui Xu (Other)
Responsible Party: Sponsor-Investigator, Guohui Xu, Principal Investigator, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2024041
Record Dates: First submitted 2024-06-22; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Unresectable Hepatocellular Carcinoma; Transarterial Chemoembolization; Camrelizumab; Apatinib
MeSH Terms: interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE plus camrelizumab and apatinib (Experimental): Procedure: TACE is performed via an injection into the hepatic artery of agents by puncturing the common femoral artery.Adriamycin(30 to 60 mg) and oxaliplatin (50-150mg) are considered as basic chemotherapy drugs in the process of transcatheter endovascular perfusion. The dose of lipiodol (5-20ml) and other embolic agent( blank microspheres/ PVA/gelatin sponge particles) were determined by diameter and blood supply type of HCC.
  Camrelizumab+apatinib: camrelizumab 200mg intravenously every 3 weeks and apatinib 250 mg orally once daily.
  Interventions: Combination Product: TACE plus camrelizumab and apatinib
- Camrelizumab plus apatinib (Active Comparator): Camrelizumab+apatinib: camrelizumab 200mg intravenously every 3 weeks and apatinib 250 mg orally once daily.
  Interventions: Combination Product: Camrelizumab and apatinib

INTERVENTIONS:
Combination Product: TACE plus camrelizumab and apatinib — TACE plus camrelizumab and apatinib group:
  Patients who were randomized to this group, TACE is performed via an injection into the hepatic artery of agents by puncturing the common femoral artery.Adriamycin(30 to 60 mg) and oxaliplatin (50-150mg) are considered as basic chemotherapy drugs in the process of transcatheter endovascular perfusion. The dose of lipiodol (5-20ml) and other embolic agent( blank microspheres/ PVA/gelatin sponge particles) were determined by diameter and blood supply type of HCC. Within 1 week after first TACE treatment, camrelizumab 200mg intravenously every 3 weeks and apatinib 250 mg orally once daily.
  Arms: TACE plus camrelizumab and apatinib
Combination Product: Camrelizumab and apatinib — Camrelizumab and apatinib group:
  Patients who were randomized to this group, camrelizumab 200mg intravenously every 3 weeks and apatinib 250 mg orally once daily.
  Arms: Camrelizumab plus apatinib

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common cancer and the third most common cause of cancer-related death worldwide. The majority of patients with HCC are diagnosed as intermediate or advanced stage disease, and not eligible for curative treatments including transplantation, resection, and ablation. Transarterial chemoembolization (TACE) is recommended as first-line treatment for patients with intermediate-stage HCC, while it is also widely used in the unresectable HCC.

The clinical efficacy and safety in advanced HCC patients of camrelizumab plus apatinib were reported in phase 3 trial (CARES-310). Camrelizumab plus apatinib with a median progression-free survival of 5.7 months and a median overall survival of 22.1 months in advanced HCC.

This study is randomized, open-label, multicenter controlled trial; which was focused in initial BCLC-B/C HCC patients. This study aimed to compare the efficacy and safety of TACE plus programmed death-1 inhibitor (camrelizumab), and anti-angiogenic therapy (apatinib) with camrelizumab plus apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or clinically confirmed hepatocellular carcinoma
2. 18-80 years old.
3. Performance status (PS) ≤ 1 (ECOG scale).
4. Barcelona clinical liver cancer (BCLC) stage B or stage C.
5. Initial treatment of hepatocellular carcinoma.
6. According to mRECIST, there is at least one measurable lesion.
7. Child Pugh score ≤ 7.
8. Participant has sufficient organ and marrow functions.
9. Expected survival time ≥ 12 weeks.
10. For women of childbearing age or male patients whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the whole treatment period and 6 months after the last medication.
11. Sign the written informed consent, and be able to follow the visit and relevant procedures specified in the plan.

Exclusion Criteria:

1. Fibrolamellar carcinoma, sarcomatoid carcinoma, cholangiocarcinoma and other components previously confirmed by histology / cytology.
2. History of hepatic encephalopathy or liver transplantation.
3. Pleural effusion, ascites and pericardial effusion with clinical symptoms requiring drainage.
4. Tumor burden≥70%, diffuse liver cancer or tumor is not suitable for mRECIST standard evaluation.
5. Received local treatment (ablation therapy, TACE), surgery resection and radiotherapy for liver cancer before the first administration.
6. Have received systemic chemotherapy, targeted therapy or immunotherapy
7. There is a significant decrease in white blood cells and platelets in peripheral blood, severe coagulation dysfunction and can not be corrected：the neutrophil<1.5×109/L, PLT<50×109/L. The INR>2.3
8. Acute or chronic active hepatitis B or C infection, hepatitis B virus (HBV-DNA) > 10^6 copies / ml; hepatitis C virus (HCV-RNA) > 10^3 copies / ml; HBsAg and anti HCV antibody were positive at the same time.
9. There is central nervous system metastasis.
10. Bleeding of esophageal or gastric varices caused by portal hypertension occurred in the past 6 months, or severe (G3) varices were found in endoscopic examination within 3 months before the first administration, or evidence of portal hypertension (including splenomegaly found in imaging examination) was found. The researchers assessed that the risk of bleeding was high and did not receive sclerotherapy or ligation under the endoscope.
11. The previous 6-month history of arteriovenous thromboembolism, including myocardial infarction, unstable angina, cerebrovascular accident, pulmonary embolism, deep vein thrombosis or any other serious thromboembolism. The thrombus of implanted vein port or catheter source or superficial vein is stable after routine anticoagulant treatment. Prophylactic use of low-molecular-weight heparin (e.g., enoxaparin 40 mg / day) is permitted.
12. Tumor thrombus of main portal vein, or involving superior mesenteric vein at the same time.
13. Aspirin (> 325 mg / day) or other drugs known to inhibit platelet function such as dipyridamole or clopidogrel were used for 7 consecutive days within 2 weeks before the first administration.
14. For uncontrolled hypertension, systolic blood pressure > 150 mmHg or diastolic blood pressure > 100 mmHg after the best medical treatment, hypertension crisis or hypertension encephalopathy history.
15. Symptomatic congestive heart failure (New York Heart Association class II-IV). Symptomatic or poorly controlled arrhythmias. The corrected QT interval (QTc) for the history or screening of congenital long QT syndrome was more than 500 ms (calculated by Fridericia method).
16. Serious bleeding tendency or coagulation dysfunction, or undergoing thrombolysis.
17. In the past 6 months, there was a history of gastrointestinal perforation and / or fistula, a history of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive enterotomy (partial colectomy or extensive enterotomy with chronic diarrhea), Crohn's disease, ulcerative colitis or long-term chronic diarrhea.
18. Previous and current pulmonary fibrosis history, interstitial pneumonia, pneumoconiosis, drug-related pneumonia, severe impairment of lung function and other lung diseases.
19. Active tuberculosis (TB), who is receiving anti TB treatment or has received anti TB treatment within one year before the first administration.
20. People with HIV infection (HIV 1 / 2 antibody positive) and known syphilis infection. Serious infection in active stage or poor clinical control.
21. Severe infection within 4 weeks before the first administration, including but not limited to hospitalization due to complications of infection, bacteremia or severe pneumonia.
22. Active autoimmune diseases requiring systemic treatment (such as the use of disease alleviation drugs, corticosteroids or immunosuppressants) occurred within 2 years before the first administration. Alternative therapies (e.g. thyroxine, insulin, or physiological corticosteroids for adrenal or pituitary insufficiency) are permitted. Known history of primary immunodeficiency. Only the patients with positive autoimmune antibody need to confirm whether there is autoimmune disease according to the judgment of researchers.
23. Immunosuppressive drugs were used within 4 weeks before the first administration, excluding local glucocorticoids or systemic glucocorticoids (i.e.

    no more than 10 Mg / day prednisone or the equivalent dose of other glucocorticoids), allowing temporary use of glucocorticoids due to dyspnea symptoms in the treatment of asthma, chronic obstructive pulmonary disease and other diseases.
24. Receive live attenuated vaccine within 4 weeks before the first administration or during the study period.
25. Major surgical procedures (craniotomy, thoracotomy or open hand) were performed within 4 weeks before the first administration (surgery) or an unhealed wound, ulcer, or fracture.
26. Uncontrolled / uncorrectable metabolic disorder or other non- malignant organ disease or systemic disease or cancer secondary reaction, which may lead to higher medical risk and / or uncertainty of survival evaluation.
27. Known to be allergic to any PD-1 monoclonal antibody component.
28. Women of childbearing age who are unwilling or unable to use acceptable methods of contraception during the whole treatment period of this trial and within 12 weeks after the last administration of the study drug (women of childbearing age include: any women who have had menarche, and have not undergone successful artificial sterilization (hysterectomy, bilateral tubal ligation, or bilateral ovariectomy), pregnancy or lactation Women; women with positive pregnancy test results at the time of inclusion or before study drug administration; If the partner is a woman of childbearing age, the subject is a fertile male without effective contraceptive measures.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | Up to 24 months, from date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Progression free survival period refers to the period from the beginning of treatment to the time when patients with cancer progress is observed or death occurs for any reason.

SECONDARY OUTCOMES:
objective response rate (ORR) | within 1 year
  The proportion of patients whose tumor volume reduction reaches the predetermined value and can maintain the minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR). That is, ORR
  * CR + PR minimum time limit. It is the sum of the proportion of complete response (CR) and partial response(PR). That is, ORR
  * CR + PR
disease control rate (DCR) | within 1 year
  It is the sum of the proportion of complete response (CR), partial response(PR) and stable disease(SD). That is, DCR
  = CR + PR + SD
overall survival (OS) | From date of randomization until the date of study completion or date of death from any cause, whichever came first, assessed up to 48 months
  the time from the beginning of treatment to death caused by any reason (the last follow-up time is for the patients who lost the visit; the end of the study is for the patients who are still alive)

CONTACTS AND LOCATIONS:
Overall Officials: Guohui Xu, Study Chair — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital and Research Institute, Chengdu, Sichuan, China